CLINICAL TRIAL: NCT04102644
Title: Limiting Adverse Birth Outcomes in Resource-Limited Settings - The LABOR Study
Brief Title: Limiting Adverse Birth Outcomes in Resource-Limited Settings
Acronym: LABOR
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0765; Z 31902 (Other: UNC)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-02

CONDITIONS: Birth Outcomes; Labor and Delivery; Respiratory Infection
Keywords: Labor and Delivery; Childbirth in limited resource setting
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women: Up to 15,000 pregnant women and their fetuses/newborns (including a pilot phase of up to 500 participant pairs)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Documentation of course and outcome of hospitalization, labor, delivery, and postpartum period

SUMMARY:
The primary objective of this research is to exhaustively document the course and outcomes of hospitalization, labor, delivery, and early postpartum course of up to 15,000 mother-newborn pairs in settings where the occurrence of adverse outcomes is high. The Investigators will gather detailed laboratory, physiologic, and clinical information, and precisely characterize major adverse diagnoses and outcomes. The resulting high-quality, granular, and generalizable data will be used to develop new algorithms to signal actionable intrapartum diagnoses and prospectively stratify women according to their risk for adverse maternal and neonatal outcomes.

DETAILED DESCRIPTION:
This is a prospective multi-country cohort study of up to 15,000 women admitted to the hospital for delivery or for management of respiratory infection. Women will be recruited and screened for study participation at the time of presentation to the hospital. Participants will be assessed through hospitalization, labor, delivery, and discharge and at 1- and 6-week postpartum contacts. Liveborn infants will be enrolled at birth and followed through 42 days of life. The pilot phase of this protocol will enroll up to 500 women in labor and their newborns and follow them through labor, delivery, and 42 days postpartum.

ELIGIBILITY:
Inclusion Criteria for women enrolled:

* Maternal age of majority
* Intrauterine singleton pregnancy
* Admission to the hospital for ANY of the following:

  1. vaginal delivery
  2. cesarean delivery in the presence of signs/symptoms of parturition, elevated blood pressure, or fever
  3. management of respiratory infection*
* Ability and willingness to provide written informed consent
* Willingness to adhere to study procedures
* Willingness to provide locator information for follow-up

  * Inclusion of participants admitted to hospital for management of respiratory infection applicable to Zambia site only.

Exclusion Criteria for women enrolled:

* Admission to the hospital for cesarean delivery in the absence of signs/symptoms of parturition, elevated blood pressure, or fever
* Any condition (social or medical) that, in the opinion of study staff, would make participation unsafe or not feasible. Study staff may note physical, psychological, or social conditions that are not explicitly stated in the eligibility criteria that could make some women poor candidates for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women and their fetuses/newborns at the Women and Newborn Hospital of the University Teaching Hospital in Lusaka, Zambia; Korle-bu Teaching Hospital in Accra, Ghana; Jawaharlal Nehru Medical College Women's and Children's Health Research Unit, KLE Academy of Higher Education and Research in Belagavi, Karnataka India; and Fakir Mohan Medical College and Hospital in Balasore, Odisha, India.
Sampling Method: Probability Sample
Enrollment: 12020 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Number of cases of maternal death or severe morbidity | enrollment - 42 days postpartum
  Maternal composite: The combined number of maternal death or incident severe morbidity arising from hemorrhage, hypertension, or infection
Number of cases of neonatal death or severe morbidity | enrollment - 42 days postpartum
  Fetal/Neonatal Composite: The combined number of Intrapartum stillbirths, neonatal deaths, neonatal encephalopathy, or neonatal sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Stringer, MD, FACOG, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- Korle Bu Teaching Hospital,, Accra, Ghana
- India (2):
  - Jawaharlal Nehru Medical College Women's and Children's Health Research Unit, KLE Academy of Higher Education and Research, Belagavi, Karnataka
  - Fakir Mohan Medical College and Hospital, Balasore, Odisha
- Women and Newborn Hospital at University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that support the study results will be shared within 6 months of the publication of primary results. As this is a multi-country study with data sharing governed by multiple research ethics and governmental oversight entities, data sharing will be subject to each country providing individual approval in accordance with its own local regulatory requirements.
Supporting Information: Study Protocol
Time Frame: Deidentified individual data that supports the study results will be shared within 6 months of the publication of primary results.
Access Criteria: See plan description

REFERENCES:
- [Derived] Walter JR, Xu S, Rogers JA. From lab to life: how wearable devices can improve health equity. Nat Commun. 2024 Jan 2;15(1):123. doi: 10.1038/s41467-023-44634-9. PMID 38167483